CLINICAL TRIAL: NCT05244382
Title: OveRCoME: functiOnal Recovery Cancer MEtastasis
Brief Title: Overcome, a Program of Therapeutic Exercise and Functional Recovery to Improve the Functional Capacity of Women With Breast Cancer and Bone Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Mario Lozano-Lozano, Principal investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Overcome project
Record Dates: First submitted 2021-12-28; First posted 2022-02-17 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Breast Neoplasm Female; Neoplasm Metastasis; Spinal Neoplasms
MeSH Terms: conditions — Neoplasm Metastasis; Spinal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Overcome group (Experimental): Three-month multimodal program. Aerobic exercise will be combined with the use of TRAG (AlterG® Anti-Gravity Treadmill®), functional recovery of motor control with feedback ultrasound and occupational therapy.
  Interventions: Other: Overcome
- Usual treatment (No Intervention): Usual medical treatment for the same period of time

INTERVENTIONS:
Other: Overcome — Multimodal program individualized and supervised 12 weeks duration (three months), with two sessions weekly face-to-face. This program will combine aerobic exercise in unloading through the use of the TRAG (AlterG® Anti-Gravity Treadmill®), functional recovery of motor control with feedback ultrasound and occupational therapy. Physical activity will be measured in parallel with the test. Likewise, the patients will be monitored by means of a heart rate sensor.
  Arms: Overcome group

SUMMARY:
The research to be carried out is aimed at patients with metastatic breast cancer, specifically bone metastases. These patients will be recruited from two hospitals in Granada, provided they meet the established inclusion criteria. With this study, it is pretend to demonstrate the benefits of a program of therapeutic exercise and functional recovery of motor control with ultrasound feedback for the improvement of the functional capacity of the women eligible to participate in the study, as well as a positive impact on the quality of life of the patients other than their survival. The effect of the Overcome program will be compared with the usual treatment in this type of pathology. To do this, a pre-intervention evaluation and another at the end of the evaluation of the variables to be measured, such as functional capacity, will be carried out. In addition other evaluation will be carried out, after 6 months to assess the long-term effects.

In addition to the three main variables such as functional capacity and quality of life, another relationship of secondary variables will be studied, such as physical state, body composition or pain threshold, among others. This study in its entirety will be carried out by the "Oncology Patient Support Unit - Take Care" in the hands of a multidisciplinary team, carrying out the intervention protocolized by physiotherapists and occupational therapists.

ELIGIBILITY:
Inclusion Criteria:

1. Having breast cancer controlled primary and occurrence of one or more bone lesions (metastases osteoblastic) with location in the pelvis, lumbar spine and / or thoracic, attributable to breast cancer
2. The bone metastasis is located only at bone level (low neurological risk).
3. Not having exercised regular physical during last 3 months.
4. ECOG (Eastern Cooperative Oncology Group) ≤ 1.
5. > 4 weeks from a major surgery and full recovery.

Exclusion Criteria:

1. Present cardiac toxicity secondary to treatments with decreased LVEF (If the LVEF percentage falls ≥ 10 points with respect to baseline or LVEF is below 50%) or QT prolongation
2. Present any other toxicity greater than grade 2 in related to the treatments you are receiving or received in advance.
3. Have spinal cord involvement, epidural involvement or instrumentation due to disease metastatic. (Moderate-high neurological risk)
4. Have started or changed treatment hormonal during the last 3 months at recruitment.
5. Present any pathology that prevents participation in a physical exercise program (PARQ-YOU).
6. Present brain metastasis.
7. Present uncontrolled hypertension (during recruitment, ≥2 / 3 evaluations <160/90 regardless of whether a regimen of antihypertensive therapy or not).
8. Having had a serious cardiovascular event recently (in the last 12 months), including, but not limited to ischemic attack transient (TIA), cerebrovascular accident (CVA) or myocardial infarction (MI).
9. Present a psychiatric illness, which would prevent the patient from signing the informed consent or adhere to the study protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 58 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | Participants will be followed over 14 weeks
  6-minute walking test
Quality of life (QLQ) | Participants will be followed over 14 weeks
  QLQ-C30 (Quality of Life of Cancer Patients) by the "European organization for reseach and treatment of cáncer quality life" (EORTC). This scale has 30 items, divided into a global health scale, 5 function subscales and 9 items/symptom scales. The scoring is obtained from through an Excel template.

SECONDARY OUTCOMES:
hand strength | Participants will be followed over 14 weeks
  Hand dynamometry, for which a digital dynamometer (TKK) 5101 Grip-D; Takey, Tokyo, Japan)
Lower limb strength | Participants will be followed over 14 weeks
  sit-up text
Body composition | Participants will be followed over 14 weeks
  Height will be measured (cm). Weight (kg), body mass index, skeletal muscle mass, and body fat percentage will be obtained using bioelectrical impedance analysis (InBody 720; Biospace, Seoul, South Korea)
Muscle architecture of multifidus muscle | Participants will be followed over 14 weeks
  Muscle ultrasound and quantitative elastosonography will be performed of the multifidus muscle. We will obtain information in real time on the parameters related to the structural organization of the tissues (normal or abnormal elasticity) with respect to the adjacent tissue.
  of the multifidus muscle.
Pain threshold on pressure, by algometry | Participants will be followed over 14 weeks
  Electronic algometer (Somedic AB, Farsta, Sweden)
Anxiety and depression | Participants will be followed over 14 weeks
  "Hospital Anxiety and Depression Scale" (HADS). Composed of two subscales: Depression and Anxiety, each with seven items. The score of each subscale can vary between 0 and 21, since each item presents four response options, ranging from absence/minimal presence = 0, to maximum presence = 3.
Opioid consumption and pain | Participants will be followed over 14 weeks
  By the scale"Brief Pain Inventory-SF". This questionnaire consists of 15 items of which only two subscales are scored organized into mean pain intensity (items 3-6) and mean pain interference (items 9A-9G), the rest of the items do not score.
Specific quality of life of the patient with bone metastasis | Participants will be followed over 14 weeks
  QLQ-BM22 (quality of life questionnaire for bone metastases) by the "European organization for reseach and treatment of cáncer quality life" (EORTC). This questionnaire consists of 22 questions, which represent eight sections on symptom scales: five identify the painful sites, and three describe the characteristics of the pain; 14 headings represent functional scales: eight, of functional interferences, and six, refer to psychosocial aspects.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Granada, Spain